CLINICAL TRIAL: NCT01161563
Title: Randomized Crossover Trial to Assess the Tolerability of GnRH Analogue Administration in Patients With Advanced Prostate Cancer
Brief Title: Randomized Crossover Trial to Assess the Tolerability of Gonadotropin Releasing Hormone (GnRH) Analogue Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TRE1001
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Results first posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Prostate Cancer
Keywords: palliative treatment; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leuprolide acetate (Active Comparator): Polymeric matrix formulation of leuprolide acetate (Eligard 45 mg) injected subcutaneously in upper or mid-abdominal area. Injection occurred either 6 months before or 6 months after injection of triptorelin pamoate suspension (Trelstar 22.5 mg) intramuscularly in the buttock.
  Interventions: Drug: Leuprolide acetate
- Triptorelin pamoate (Active Comparator): Triptorelin pamoate suspension (Trelstar 22.5 mg) injected intramuscularly in the buttock. Injection occurred either 6 months before or 6 months after injection of polymeric matrix formulation of leuprolide acetate (Eligard 45 mg) subcutaneously in upper or mid-abdominal area.
  Interventions: Drug: Triptorelin pamoate

INTERVENTIONS:
Drug: Triptorelin pamoate — Triptorelin pamoate for injectable suspension 22.5 mg administered as a single intramuscular injection in either buttock
  Arms: Triptorelin pamoate
Drug: Leuprolide acetate — Leuprolide acetate for injectable suspension 45 mg administered as a single subcutaneous injection in the upper- or mid-abdominal area.
  Arms: Leuprolide acetate

SUMMARY:
The purpose of this study is to compare how subjects feel after receiving injections of two different types of GnRH six months apart. One injection is given under the skin of the abdomen, and the other one into the muscle of the buttock or thigh.

DETAILED DESCRIPTION:
GnRH is given as an injection. Injections of GnRH can be uncomfortable, causing a feeling of burning or stinging. The uncomfortable feeling may be caused by differences in the types of GnRH and the site of the injection (under the skin of the abdomen, or into the muscle of the buttock or thigh).

ELIGIBILITY:
Inclusion Criteria:

* Male patients with a diagnosis of advanced prostate cancer for whom treatment with triptorelin pamoate or leuprolide acetate is indicated;
* At least 18 years of age;
* Life expectancy of at least 1 year;
* Capable of completing the study questionnaires without assistance.

Exclusion Criteria:

* Patients for whom treatment with triptorelin pamoate or leuprolide acetate is contraindicated;
* Known hypersensitivity to triptorelin, leuprolide or any other GnRH or luteinizing hormone releasing hormone (LHRH) agonists, or GnRH or LHRH;
* Clinically significant systemic disease or condition that would, in the investigator's opinion, lead to undue risk following administration of either triptorelin or leuprolide;
* History of alcohol/drug abuse within the past year;
* History of significant medical problems that may confound the outcome of this study;
* Requires concomitant medications that may affect study assessments (e.g., topical medications used for pretreatment of injection site pain);
* Participated in another investigational drug study within 30 days
* Judged by the investigator to be unsuitable for enrollment in this study for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn McIlwain, BS, Study Director — Watson Pharmaceuticals, Inc.
Locations (16):
- United States (16):
  - Watson Investigational Site, Homewood, Alabama
  - Watson Investigational Site, Daytona Beach, Florida
  - Watson Investigational Site, Orange City, Florida
  - Watson Investigational Site, Coeur d'Alene, Idaho
  - Watson Investigational Site, Carmel, Indiana
  - Watson Investigational Site, Jeffersonville, Indiana
  - Watson Investigational Site, Shreveport, Louisiana
  - Watson Investigational Site, Las Vegas, Nevada
  - Watson Investigational Site, Mount Laurel, New Jersey
  - Watson Investigational Site, Voorhees Township, New Jersey
  - Watson Investigational Site, Albany, New York
  - Watson Investigational Site, Syracuse, New York
  - Watson Investigational Site, Lancaster, Pennsylvania
  - Watson Investigational Site, Myrtle Beach, South Carolina
  - Watson Investigational Site, Dallas, Texas
  - Watson Investigational Site, Norfolk, Virginia

REFERENCES:
- [Derived] Shore ND, Sieber P, Schimke L, Perzin A, Olsen S. Comparison of tolerability and adverse events following treatment with two GnRH agonists in patients with advanced prostate cancer. Urol Nurs. 2013 Sep-Oct;33(5):236-44, 248. PMID 24354113

RESULTS

PARTICIPANT FLOW:
Groups:
- Triptorelin First, Then Leuprolide Acetate: Injection of triptorelin pamoate suspension (Trelstar 22.5 mg) intramuscularly in the buttock, followed 6 months later by injection of polymeric matrix formulation of leuprolide acetate (Eligard 45 mg) in the upper or mid-abdominal area.
  A detailed breakdown of participant flow by treatment period for each arm is not available.
- Leuprolide Acetate First, Then Triptorelin: Injection of polymeric matrix formulation of leuprolide acetate (Eligard 45 mg) in the upper or mid-abdominal area, followed 6 months later by injection of triptorelin pamoate suspension (Trelstar 22.5 mg) intramuscularly in the buttock.
  A detailed breakdown of participant flow by treatment period for each arm is not available.
Period: Overall Study
Arm/Group | Triptorelin First, Then Leuprolide Acetate | Leuprolide Acetate First, Then Triptorelin
Started | 63 | 55
Completed | 58 | 49
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Leuprolide Acetate First, Then Triptorelin: Polymeric matrix formulation of leuprolide acetate (Eligard 45 mg) injected subcutaneously in upper or mid-abdominal area 6 months before injection of triptorelin pamoate suspension (Trelstar 22.5 mg) intramuscularly in the buttock.
- Triptorelin First, Then Leuprolide Acetate: Triptorelin pamoate suspension (Trelstar 22.5 mg) injected intramuscularly in the buttock 6 months before injection of polymeric matrix formulation of leuprolide acetate (Eligard 45 mg) subcutaneously in upper or mid-abdominal area.
- Total: Total of all reporting groups
Arm/Group | Leuprolide Acetate First, Then Triptorelin | Triptorelin First, Then Leuprolide Acetate | Total
Number analyzed (Participants) | 55 | 63 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 29
  >=65 years | 43 | 46 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 75.0 (9.6) | 73.2 (9.6) | 74 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 55 | 63 | 118
Region of Enrollment [Number; unit: participants]
  United States | 55 | 63 | 118

OUTCOME MEASURES:

1. Primary Outcome: Patient Bother From Injection Site Burning and/or Stinging
Description: Questionnaire responses recorded on a Visual Analog Scale (VAS), which has a range of 0-100 mm, assessed approximately 15 minutes post-injection
Time Frame: 15 minutes
Population: Per-protocol population, defined as all patients who receive both study drugs and complete both post-injection questionnaires.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Leuprolide Acetate: Results combined for the leuprolide acetate treatment period for both randomization groups for the Per-protocol population (n=107), defined as all patients who receive both study drugs and complete both post-injection questionnaires.
- Triptorelin Pamoate: Results combined for the triptorelin pamoate treatment period for both randomization groups for the Per-protocol population (n=107), defined as all patients who receive both study drugs and complete both post-injection questionnaires.
Arm/Group | Leuprolide Acetate | Triptorelin Pamoate
Number analyzed (Participants) | 107 | 107
units on a scale | 23.87 [19.98 to 27.76] | 5.84 [1.95 to 9.73]

2. Secondary Outcome: Discomfort From Injection
Description: as for outcome 1
Time Frame: 15 minutes
Population: Per-protocol population, defined as all subjects who receive both study drugs and complete both post-injection questionnaires.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Leuprolide Acetate | Triptorelin Pamoate
Number analyzed (Participants) | 107 | 107
units on a scale | 20.53 [16.49 to 24.56] | 5.88 [1.85 to 9.92]

ADVERSE EVENTS:
Arm/Group | Leuprolide Acetate | Triptorelin Pamoate
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/118
Other Adverse Events (participants affected / at risk) | 0/118 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less